CLINICAL TRIAL: NCT01502059
Title: The Effectiveness of Pilates to Treat Low Back Pain: A Randomized Controlled Trial
Brief Title: Pilates to Treat Low Back Pain
Acronym: PTLBP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Anamaria Jones, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP UNIFESP 0208/11
Record Dates: First submitted 2011-12-27; First posted 2011-12-30 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Pain; Quality of Life
Keywords: Pilates; Exercise; Treatment; Low back pain; Pain; Function
MeSH Terms: conditions — Pain; Motor Activity; Low Back Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilates Group (Experimental): This group keep their usual treatment and did a Pilates treatment twice a week (one hour each class) during 90 days.
  Interventions: Other: Pilates
- Control Groups (No Intervention): This group keep their usual treatment and can do the Pilates training after the end of the study.

INTERVENTIONS:
Other: Pilates — Pilates training - twice a week (one hour per class) during 90 days
  Arms: Pilates Group

SUMMARY:
This is a randomized controlled trial, with blinded assessor to evaluate the effectiveness of Pilates to treat low back pain.

Hypothesis - the Pilates group will have best results than the control group (usual medicament treatment).

DETAILED DESCRIPTION:
Background:

Low back pain (LBP) is a common problem among adults. Approximately 70-85% of the adult population experiences this painful complaint at some point in their lives, making LBP the second most common reason for a visit to a clinician. Despite the frequency of this diagnosis, conventional treatment does not always provide patients the desired results of reduced pain and return of normal function. For these patients, alternative modalities are available to assist in the control of pain. These options include chiropractic care, physical therapy, massage therapy, and modalities that fall under the auspices of complementary and alternative medicine, such as acupuncture. Unfortunately, Clinical trials evaluating the efficacy of a variety of interventions for chronic non-specific low back pain indicate limited effectiveness for most commonly applied interventions and approaches.

Objectives:

To evaluate the effectiveness of a mat and studio Pilates program on pain, function, quality of life and NHAI consumption for chronic non-specific low back pain patients.

Methods:

Eligible patient include: chronic non-specific low back pain; age between 18 and 65 years; pain ranging from 4 to 8 in a numerical pain scale. Patients with previous surgery, other causes of low back pain, fibromyalgia, regular physical activity (three or more times per week for at least three months); labor lawsuit and body mass index more than 30. Sixty patients were randomized to the Experimental Group (EG) or Control Group (CG). Patients in EG participated in 90 days of mat and studio Pilates program twice a week (50 minutes per class) and the CG remained with their usual medicament treatment and were included in a waiting list for physiotherapy. Assessment for pain (VAS), function (Roland Morris questionnaire), quality of life (SF-36) and NHAI consumption were done at baseline, after 45 days (T45), after 90 days (T90 - end of the program), after 90 days (T180 - follow up) by a blinded assessor.

ELIGIBILITY:
Inclusion Criteria:

* non specific mechanical low back pain
* visual analogue scale for pain ranging from 4 to 7

Exclusion Criteria:

* previous back surgery
* spinal tumor
* spinal fracture
* pregnancy
* fibromyalgia
* inflammatory or infectious spinal diseases
* litigant patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in pain | Baseline, after 45, 90 and 180 days
  Measured with the visual analogue scale ranging from 0 to 10

SECONDARY OUTCOMES:
Change in function | Baseline, after 45, 90 and 180 days
  Measured by the questionnaire Roland Morris
Change in quality of life | Baseline, after 45, 90 and 180 days
  Measured by the SF-36 questionnaire
Change in nonsteroidal antiinflammatory drugs (NSAIDs) consumption | Baseline, after 45, 90 and 180 days
  Measured by counting the number of tablets consumed per month

CONTACTS AND LOCATIONS:
Overall Officials: Anamaria Jones, PT, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil